CLINICAL TRIAL: NCT04548401
Title: Effect of Antiplatelet Therapy on Cognition After Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hai-Bin Shi, Professor, Nanjing Medical University
Other Study IDs: aSAH016
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antiplatelet-N group: Patients with ruptured aneurysm underwent coiling alone, without post-treatment antiplatelet therapy
- Antiplatelet-Y group: Patients with ruptured aneurysm underwent stent assisted coiling, with post-treatment antiplatelet therapy (aspirin and/or clopidogrel or ticagrelor)
  Interventions: Drug: Antiplatelet Drug

INTERVENTIONS:
Drug: Antiplatelet Drug — aspirin and/or clopidogrel or ticagrelor
  Groups: Antiplatelet-Y group

SUMMARY:
Deficits in memory, executive function, and language are common cognitive sequelae of aneurysmal subarachnoid hemorrhage (aSAH). Previous study demonstrated that post-treatment antiplatelet therapy reduced risk for delayed cerebral ischemia caused by aSAH. However, the effect of antiplatelet therapy on cognition after aSAH is unclear. The aim of this study was to assess the effect of antiplatelet therapy on cognition after aSAH.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with SAH in whom the aneurysm was proven by conventional angiography; 2. Baseline Hunt-Hess grade I-III; 3. patients received endovascular treatment

Exclusion Criteria:

* 1. Hunt-Hess grade IV-V; 2. Non-aneurysmal SAH; 3. Dementia in other diseases; 4. Lacking of 6-8 month MoCA evaluation.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with aSAH who received endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) Test | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Hai Bin Shi, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided